CLINICAL TRIAL: NCT04695990
Title: Study on the Clinical and Mechanism of Wenyang Huoxue Decoction in Treating Heart Failure After Myocardial Infarction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jun Li (Other)
Responsible Party: Sponsor-Investigator, Jun Li, Chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: wyhx-2020
Record Dates: First submitted 2020-11-29; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure; Myocardial Infarction
Keywords: Wenyang Huoxue decoction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): On the basis of basic western medicine treatment (secondary prevention of coronary heart disease + anti-heart failure treatment), Patients in this group will be given Wenyang Huoxue Decoction, one dose per day, administered in two doses, 150-200 mL each time, for 12 weeks.
  Interventions: Drug: Wenyang Huoxue Decoction
- Control group (Placebo Comparator): On the basis of basic western medicine treatment (secondary prevention of coronary heart disease + anti-heart failure treatment), Patients in this group will be given placebo, one dose per day, administered in two doses, 150-200 mL each time, for 12 weeks.
  Interventions: Drug: Wenyang Huoxue placebo

INTERVENTIONS:
Drug: Wenyang Huoxue Decoction — Wenyang Huoxue granules
  Other Names: WYHX
  Arms: Experimental group
Drug: Wenyang Huoxue placebo — Wenyang Huoxue placebo have an identical appearance and scent as the active treatment granules.
  Other Names: WYHX placebo
  Arms: Control group

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel clinical trial in a Chinese population with heart failure after myocardial infarction. The objective is to observe the efficacy and safety of Wenyang huoxue fang in the treatment of heart failure after myocardial infarction.

DETAILED DESCRIPTION:
Currently, there is a lack of high-quality evidence-based support for TCM treatment of heart failure after myocardial infarction. In addition, previous studies have found that the method of warming Yang and activating blood circulation is effective in treating coronary heart disease, and the core pathogenesis of heart failure after myocardial infarction is also Yang deficiency and blood stasis. Therefore, this project aims to evaluate the clinical value of warming Yang and activating blood circulation in the treatment of heart failure after myocardial infarction. Through pharmacological research and detection, the efficacy of Wenyang huoxue prescription in heart failure rats after intervention of myocardial infarction was evaluated, mir-233-ISO signaling pathway was detected before and after treatment, and its mechanism of action was further clarified from the perspective of epigenetics and classical pathway of heart failure.

Objective To investigate the efficacy and safety of Wenyang Huoxue fang in the treatment of heart failure after myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* A history of acute myocardial infarction;
* Cardiac function grade II-IV;
* LVEF 40% or less; NT-proBNP level ≥ 450 pg/mL; -All men and women can sign the informed consent form.-

Exclusion Criteria:

* Coronary artery bypass grafting was performed within 12 weeks.
* Undergo or possibly undergo cardiac resynchronization therapy;
* Primary valvular disease, left ventricular outflow tract obstruction, myocarditis, aneurysm, uncontrolled severe arrhythmia, cardiogenic shock, unstable angina pectoris, or acute myocardial infarction;
* Having a serious primary liver, kidney or blood system disease or having a serious mental illness or a systemic disease that is out of control;
* Serum creatinine > 194.5 mol/L or serum potassium > 5.5mmol /L;
* The level of alanine aminotransferase or alkaline phosphatase is 1.5 times of the normal upper limit ;
* Abnormal blood pressure control, systolic blood pressure exceeding 180mmHg or diastolic blood pressure exceeding 110mmHg;
* Pregnancy or lactation;
* Known or suspected allergy to research drugs;
* To receive another investigational drug within 30 days of randomization or to be unwilling or unable to provide written consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular events | One months to 1 year after drug intervention
  The number of major cardiovascular events，These include death, myocardial infarction, and rehospitalization

SECONDARY OUTCOMES:
Main observation indicators | Into the group day 1, week 4, week 8, week 12
  The numerical of NT-proBNP
Secondary observation index | Into the group day 1, week 4, week 8, week 12
  The Left ventricular ejection fractione of chocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Result] Hildebrandt P. Systolic and nonsystolic heart failure: equally serious threats. JAMA. 2006 Nov 8;296(18):2259-60. doi: 10.1001/jama.296.18.2259. No abstract available. PMID 17090774
- [Result] Gheorghiade M, Bonow RO. Chronic heart failure in the United States: a manifestation of coronary artery disease. Circulation. 1998 Jan 27;97(3):282-9. doi: 10.1161/01.cir.97.3.282. No abstract available. PMID 9462531
- [Result] Gerber Y, Melton LJ 3rd, Weston SA, Roger VL. Association between myocardial infarction and fractures: an emerging phenomenon. Circulation. 2011 Jul 19;124(3):297-303. doi: 10.1161/CIRCULATIONAHA.110.007195. Epub 2011 Jun 27. PMID 21709062
- [Result] Ezekowitz JA, Kaul P, Bakal JA, Armstrong PW, Welsh RC, McAlister FA. Declining in-hospital mortality and increasing heart failure incidence in elderly patients with first myocardial infarction. J Am Coll Cardiol. 2009 Jan 6;53(1):13-20. doi: 10.1016/j.jacc.2008.08.067. PMID 19118718